CLINICAL TRIAL: NCT05396937
Title: Efficacy and Safety of Multifocal Stereotactic Radiotherapy Combined With Atezolizumab and Bevacizumab in the Treatment of Metastatic Hepatocellular Carcinoma: An Open-label, Single-arm Exploratory Study
Brief Title: Efficacy and Safety of T+A+RAD in HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-RAD
Record Dates: First submitted 2022-04-02; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T+A+RAD (Experimental)
  Interventions: Radiation: Multifocal Stereotactic Radiotherapy; Drug: Atezolizumab Injection [Tecentriq]; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Multifocal Stereotactic Radiotherapy — Radiotherapy will be given in combination with atezolizumab and bevacizumab. The patient will be initially treated with atezolizumab and bevacizumab after enrollment. Radiotherapy will be administered to the metastases 1-2 weeks after the completion of the first intravenous injection of atezolizumab and bevacizumab, in the mode of multifocal stereotactic radiotherapy, with a planned total dose to the planned target volume of 25-50 Gy in five divided doses of 5-10 Gy/fraction. Systemic therapy could be continued 48 hours after completion of radiotherapy.
Drug: Atezolizumab Injection [Tecentriq] — Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21 day cycle
Drug: Bevacizumab — Bevacizumab will be administered by IV, 10 mg/kg on day 1 of each 21 day cycle

SUMMARY:
This is An Open-label, Single-arm Exploratory Study to determine the efficacy and safety of Multifocal Stereotactic Radiotherapy Combined with Atezolizumab and Bevacizumab in the Treatment of Metastatic Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female between the ages of 18 and 70;
2. signed informed consent;
3. The researchers believe that patients have the ability to comply with the research program;
4. hepatocellular carcinoma (HCC) by histological or cytological or clinical diagnosis;
5. imaging examination confirmed extrahepatic dissemination, including at least one evaluable (according to the criteria of RECIST1.1) extrahepatic metastasis;
6. disease is not suitable for radical surgery;
7. Patients who have not received radiotherapy or treatment with aletirizumab and/or bevacizumab;
8. Early treatment allows tyrosine kinase inhibitors (TKI) treatment or immunotherapy;
9. Pre-treatment tumor tissue samples (if available); If tumor tissue is available, submit 1 formalin-fixed, paraffin embedded (FFPE) tumor sample from a paraffin block (preferred) or approximately 10-15 slides containing unstained, off-the-shelf, serial sections together with a pathology report within 4 weeks of enrollment. If the FFPE samples described above are not available, samples of any type (including fine needle aspiration biopsy samples, cell mass samples [e.g., samples from pleural effusion], and irrigation samples) may also be accepted. A relevant pathology report shall be provided with the sample. If tumor tissue is not available (e.g., exhausted for previous diagnostic tests), the patient remains eligible to participate;
10. ECOG performance status of 0 or 1 within 14 days before enrollment;
11. Child-Pugh A or ≤ 7 grade B within 14 days before enrollment;
12. sufficient hematology and organ function, based on the results of the following laboratory tests obtained within 14 days before enrollment (unless otherwise specified): absolute neutropcount (ANC) ≥ 1.5 × 109/L (1500/μL), without granulocyte colony-stimulating factor support; lymphocyte count ≥ 0.5 × 109/L (500/μL); platelet count ≥ 75 × 109/L (75, 000/μL) or ≥ 60 × 109/L (60, 000/μL) but normal prothrombin time without blood transfusion; hemoglobin ≥ 90 g/L (9 g/dL), in order to meet this criterion, Patients may be allowed to have blood transfusions; AST, ALT and alkaline phosphatase (ALT) ≤ 5 times the upper limit of the normal value; Serum bilirubin ≤ 3 times the upper limit of the normal value; Serum creatinine ≤ 1.5 times the upper limit of normal value or calculated creatinine clearance ≥ 50 mL/min (calculated using Cockcroft-Gault formula); Serum albumin ≥ 28 g/L (2.8 g/dL) Urine cellulose strip test results in proteinuria < 2 + (performed within 14 days prior to starting study treatment); patients with baseline cellulose strip test results of ≥ 2 + proteinuria should collect 24 hours of urine and then must demonstrate < 1g of urine protein in 24 hours.
13. Any acute, clinically significant treatment-related toxicity (caused by previous treatment) must have been alleviated to ≤ 1 grade before entering the study, except hair loss;
14. HIV antibody test results were negative at the time of screening;
15. Patients with active hepatitis B virus (HBV) infection: HBV DNA < 2000 IU/mL obtained within 28 days before the start of study treatment, and at least 7 days of anti-HBV treatment (according to the local standard treatment, such as entecavir) before the study and willing to continue treatment during the study
16. Women of childbearing age must have a negative pregnancy test (beta HCG) before starting treatment, women and men of reproductive age (having sex with women of reproductive age) must agree to use effective contraceptive measures during treatment and 6 months after the last dose of treatment.

Exclusion Criteria:

1. History of soft meningitis;
2. Current or previous autoimmune disease or immune deficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions: patients with autoimmune hypothyroidism and receiving thyroid hormone replacement therapy were eligible to participate in the study; patients with controlled type 1 diabetes receiving insulin therapy were eligible to participate in the study; patients with eczema, psoriasis, chronic lichen simplex, or vitiligo with dermatologic clinical manifestations only (e.g., patients with psoriasis arthritis were excluded) were eligible to participate as long as all of the following conditions were met: 1. Rash area must be < 10% of body surface area; 2. The disease was well controlled at baseline and required only low-potency topical glucocorticoids. 3. In the past 12 months, the original condition did not appear to require psoralen plus A-band ultraviolet radiation, methotrexate, vitamin A acid, biological agents, oral calcineurin inhibitors or highly active or oral corticosteroids treatment of acute exacerbation;
3. Idiopathic pulmonary fibrosis, organizing pneumonia (e.g., obliterative bronchitis), drug pneumonia or idiopathic pneumonia or evidence of active pneumonia on screening chest computed tomography (CT) scan; A history of radiation pneumonitis in the area of allowable radiation (fibrosis);
4. known active tuberculosis;
5. Significant cardiovascular disease within 3 months before the start of study treatment (for example, New York Heart Association grade II or worse heart disease, myocardial infarction or cerebrovascular accident within 3 months before the start of study treatment), unstable arrhythmia or unstable angina;
6. History of congenital long QT syndrome or corrected QT interval > 500 ms at screening (calculated using Fridericia method);
7. history of uncorrectable serum potassium, calcium or magnesium electrolyte disorders;
8. Patients who have undergone major surgery (except diagnosis) within 4 weeks before the start of study treatment or are expected to undergo major surgery during the study period;
9. Have had malignant tumors other than HCC within 5 years before screening, except for those with negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated in situ cervical cancer, non-melanoma skin cancer, localized prostate cancer, in situ cancer or stage I uterine cancer;
10. Severe infection within 4 weeks before the start of study treatment, including but not limited to hospitalization due to infection, bacteremia or severe pneumonia complications;
11. Oral or intravenous administration of therapeutic antibiotics within 2 weeks prior to the start of study treatment; Patients receiving preventive antibiotics (e.g., prevention of urinary tract infections or chronic obstructive pulmonary disease exacerbations) were eligible to participate;
12. Previous allogenic stem cell or solid organ transplantation;
13. Patients who have received live attenuated vaccine treatment within 4 weeks before the start of study treatment, or are expected to receive such vaccine during the treatment period or 5 months after the last administration of altezumab;
14. Untreated or incompletely treated patients with esophageal and/or gastric varices with bleeding or high risk of bleeding; Prior to enrollment, patients must undergo ultrasound, CT, MRI, or liver elasticity testing to assess the size of all varices (small to large) and be treated according to local standard of care. Patients who have had a corresponding examination within 6 months prior to starting study treatment do not need to repeat the examination;
15. Coinfection with HBV and HCV. Patients with a history of HCV infection and a negative PCR result for HCV RNA were considered not infected with HCV;
16. symptomatic, untreated or progressive central nervous system (CNS) metastases; Asymptomatic patients with treated CNS disease were eligible for the study if they met all of the following criteria: they had disease outside the CNS that could be measured according to RECIST v1.1; they had no history of intracranial hemorrhage or intraspinal hemorrhage; their metastatic disease was limited to the Cerebellar or supratentorial region (i.e., they had no midbrain, pontine, medullary, or spinal cord metastases); there was no evidence of progression between completing CNS-guided therapy and starting study treatment; the patients had not been treated with stereotactic, whole brain radiotherapy, and/or neurosurgical resection within 28 days prior to starting study treatment; and the patients did not have the need for ongoing glucocorticoid therapy for CNS disease. A stable dose of anticonvulsant therapy was allowed. Asymptomatic patients with newly detected CNS metastases at screening, after radiotherapy or surgery, were eligible to participate in the study without the need for repeat screening brain scans;
17. patients can not accept follow-up or are participating in other liver cancer comprehensive treatment of the relevant clinical trials;
18. The researchers believe that subjects who are not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate, ORR | through study completion, an average of 1 year
  Percentage of Participants with Objective Response According To Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Duration of Objective Response (DoR) | through study completion, an average of 1 year
  time interval between objective response to progression
Disease Control Rate (DCR) | through study completion, an average of 1 year
  CR+PR+SD
Time to progression (TTP) | through study completion
  From screening to the first occurrence of disease progression from any cause up to end of study
Progression-free survival (PFS) | through study completion
  From screening to the first occurrence of disease progression or death from any cause up to end of study
Overall survival (OS) | through study completion
  From screening to death from any cause up to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No